CLINICAL TRIAL: NCT03713463
Title: An Observational, Multicenter Study to Evaluate the Benefits of Regular Intake of Standard ONS in Indian Adults
Brief Title: Benefits of Standard ONS in Indian Adults
Status: Terminated | Type: Observational
Why Stopped: COVID-19 enrollment challenges
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: DA18
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Poor Nutrition
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oral Nutritional Supplement (ONS): 2 servings per day ONS
  Interventions: Other: Oral Nutritional Supplement (ONS)

INTERVENTIONS:
Other: Oral Nutritional Supplement (ONS) — Per standard of care (SOC)

SUMMARY:
This is a prospective, single arm, baseline-controlled multicenter study to observe benefits on Oral Nutritional Supplement (ONS) intake in adults with medical conditions associated with poor nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adult patients >or equal to 45 years of age
* Patients at the risk of malnutrition (MST > or equal to 2)
* Patients who understand nature of the study, willing to participate in all scheduled visits and trial procedures & provide a written informed consent.

Exclusion Criteria:

* Subject using commercially available macronutrient food supplements or another ONS
* History or evidence of hypersensitivity to any component of study product
* History of any Gastrointestinal disorder/surgery that affects digestion and/or absorption of food
* Evidence of active TB, Hepatitis B, Hepatitis C or HIV infection, type 1 or type 2 diabetes mellitus, malignancy and any other disease affecting appetite and weight loss
* History or evidence of any medical condition that in the opinion of Investigator can interfere with the study assessment of outcome or Patients with scheduled surgery during the duration of the study
* Subjects who are unlikely to comply with the study protocol or follow up regularly for study assessments
* Pregnant or lactating women

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out-patient healthcare clinics across India
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2020-09-06 (Actual); Study Completion 2020-09-06 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline to 12 weeks
  Measured weight kg

SECONDARY OUTCOMES:
Hand Grip | Baseline to 12 weeks
  Dynamometer
Quality of Life (QoL) | Baseline to 12 weeks
  World Health Organization QOL-BREF Questionnaire; 4 Domain scores scaled in a positive direction (very dissatisfied - very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Kadhe, MD, Study Chair — Abbott Healthcare PVT. LTD.
Locations (45):
- India (45):
  - Subramanyam's Day Care Center, Bangalore
  - Sunidhi Health Centre, Bangalore
  - Dr.Vinay J. Clinic, Bangalore
  - Sri Sai Health Care Center, Bangalore
  - Chandra Chest and Diabetes Care Center, Chennai
  - Dr. Srinivasan Clinic, Chennai
  - Vasavi Clinic, Chennai
  - Sree Narayana Nursing Home, Chennai
  - Adhiparasakthi Clinic, Chennai
  - Sow-Krish Clinic, Chennai
  - Javantika Clinic, Chennai
  - Prime Family Medical Centre, Chennai
  - Dr. U. V. Mohan Clinic, Chennai
  - Dr. S. Nagrajan Clinic, Chennai
  - Vcure Clinic, Chennai
  - Dr. Sriram V. Clinic, Chennai
  - Goel Clinic, Delhi
  - Joshi Clinic, Delhi
  - Sharma Clinic, Delhi
  - Jain Clinic, Delhi
  - Sanjeevan Clinic, Delhi
  - Dr. Asoktaru Sengupta Clinic, Howrah
  - Dr. Mridul Bera Clinic, Howrah
  - Dr. Jagdish singh Clinic, Hyderabad
  - Geetha Hospital, Hyderabad
  - Maxcure Hospitals, Hyderabad
  - City Clinic, Hyderabad
  - Healthy Lifestyle Clinic, Kolkata, Kolkata
  - Dass Medical Hall, Kolkata
  - Dr. Arabinda Halder Clinic, Kolkata
  - Dr. Parinata Roy Clinic, Kolkata
  - Dr. A. K. Chatterjee Clinic, Kolkata
  - Dr. O. P. Sharma Clinic, Kolkata
  - Qureshi Clinic, Mumbai
  - Contractor Clinic, Mumbai
  - Dhabolkar Clinic, Mumbai
  - Bhulchandani Hospital, Mumbai
  - Dr. S. Vikas Clinic, Mumbai
  - Ajitkumar Clinic, Mumbai
  - Dr. A. Mahadev Clinic, Secunderabad
  - Gayatri Clinic, Secunderabad
  - Boricha Clinic, Thane
  - Devrukhar Clinic, Thane
  - Pawar Clinic, Thane
  - Thakkar Clinic, Thane

IPD SHARING:
Plan to Share IPD: Undecided